CLINICAL TRIAL: NCT05743673
Title: A Feasibility Study of the SHAPE™ Test of Aerobic Fitness in Older Adults Presenting for Moderate to High-risk Surgery
Brief Title: SHAPE Test for Preoperative Risk Stratification
Acronym: SHAPEPAT
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Zyad Carr, Associate Professor, Department of Anesthesiology, Yale University
Other Study IDs: 2000033885
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Perioperative/Postoperative Complications; Aerobic Capacity
Keywords: perioperative risk stratification; submaximal cardiopulmonary exercise testing; postoperative complications; perioperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Validation Cohort: Older subjects (>60 years old) presenting for moderate to high-risk surgical procedure with reported subjective metabolic equivalents of >4 METS and with a score of <4 on the revised cardiac risk index (RCRI) undergoing submaximal exercise testing.
  Interventions: Device: Shape II

INTERVENTIONS:
Device: Shape II — cardiopulmonary exercise testing apparatus

SUMMARY:
Primary Objective Characterizing precise functional capacity in surgical patients is critical for risk stratification and identification of patients at high risk for perioperative complications. The primary objective for the study is to evaluate the feasibility of effective subject recruitment of an FDA-approved simplified cardiopulmonary exercise testing apparatus in adults >60 years old prior to moderate to high-risk surgery. In addition, by development of a validation cohort of older adults, defined as >60 years old, self-reporting >4 METS and with a score of <2 on the revised cardiac risk index (RCRI)1 we will compare its effectiveness when compared to conventional preoperative evaluation measures (METS determination by standard scoring and Duke Activity Status Index) to SHAPE™ testing.

DETAILED DESCRIPTION:
The submaximal heart and pulmonary evaluation (SHAPE™) test is an FDA approved cardiopulmonary exercise testing (CPET) system that provides a rapid and non-invasive way of characterizing cardiopulmonary reserve in a variety of medical conditions3,4. Traditional CPET testing has demonstrated predictive power in the assessment of postoperative mortality, hospital length of stay and other postoperative complications after lung resection, abdominal aortic aneurysm repair and liver transplants5-7. A unique advantage of SHAPE™ testing is that functional capacity variables are both obtained at rest and during sub-maximal exercise, potentially mimicking elicited conditions associated with surgical stress, as well as assist in determining the specific component of the physiological system under duress during testing (cardiac vs. pulmonary). Additionally, unlike conventional CPET, a maximum exercise effort is not required, making it an attractive option for patients with cardiopulmonary or musculoskeletal disorders and elderly patients who are unable to undergo the higher intensity exercise testing associated with traditional CPET. Finally, investigation of unique SHAPE™ variables (e.g. GXcap/Δend-tidal C02) which have been observed to be sensitive performance indicators for a variety of cardiovascular diseases such as heart failure with preserved ejection fraction, may prove more sensitive to traditional CPET variables or conventional echocardiography3.

This is a prospective, non-randomized feasibility study to evaluate the effectiveness of subject recruitment of an FDA-approved simplified cardiopulmonary exercise testing apparatus in adults >60 years old prior to moderate to high-risk surgery. Pre-screened research subjects will be approached by telephone or in-person within the pre-surgical evaluation clinic prior to their surgery. We hypothesize that >25% of eligible subjects will be recruited in the investigation. A single 35 minute in-person session will be performed where subjective metabolic equivalents will be assessed, and experimental session of the SHAPE™ medical system testing apparatus. Research subjects will then be released after survey. A follow-up telephone call at 24 hours will assess any adverse events related to the experimental session. For the period of 30 days after their scheduled surgery, minor and major postoperative complications will be extracted from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Aged >60 years
* Scheduled for pre-surgical evaluation for moderate to high-risk surgical procedure.
* RCRI <2 based on screening of preoperative co-morbidities.
* Provision of signed and dated informed consent form

Exclusion Criteria:

1. Age <60 years old
2. Subjective METS <4
3. Inability to give independent informed consent
4. Revised Cardiac Risk Index (RCRI) >2
5. Neurological impairment with motor limitations
6. Mental impairment leading to inability to cooperate
7. Recent NSTEMI or STEMI type myocardial infarction (within 6 months)
8. Angina (stable or unstable, within 6 months)
9. Uncorrected severe valvular heart disease (severe aortic, tricuspid, or mitral stenosis)
10. Recent exacerbation of congestive heart failure (requiring hospitalization, within 6 months)
11. Acute pulmonary embolism or deep vein thrombosis (within past 6 months)
12. Uncontrolled pulmonary edema
13. Uncontrolled symptomatic arrhythmias
14. Active endocarditis
15. Acute myocarditis or pericarditis
16. Active wheezing or home oxygen use
17. Recent exacerbation of chronic obstructive pulmonary disease or asthma or pneumonia (requiring hospitalization, within 6 months)
18. Inability to perform components of the SHAPE test (severe hip flexion limitation, severe osteoarthritis of knee or hip, limb immobilization, ambulation with a walker, can or crutches, baseline balance irregularities
19. Diagnosis of vertigo
20. Known allergic reactions to components of the SHAPE medical system apparatus disposable mouthpiece.
21. Active enrollment in an interventional clinical trial within the enrollment period of the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The overall goal is the development of a validation cohort of older adults, defined as >60 years old, self-reporting >4 METS and with a score of <2 on the revised cardiac risk index (RCRI)1
Sampling Method: Non-Probability Sample
Enrollment: 371 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Recruitment Success | 0-30 days
  The primary objective for the study is a study enrollment rate of 25% of eligible candidates.
  Within the parameters of a feasibility study, the following questions will also be addressed:
  * Physical capacity of clinic to handle the number of participants in the study.
  * Adequate communication and time frame to efficiently perform abbreviated cardiopulmonary exercise testing in high-volume preoperative testing environment.
  * Adequate software and hardware to capture and use data obtained from abbreviated cardiopulmonary exercise testing.
  * Determination of adequate institutional, departmental and clinical support to maintain and perform abbreviated cardiopulmonary exercise testing as an adjunct for preoperative testing.
  * Does abbreviated cardiopulmonary testing in a preoperative testing environment improve access to care in a diverse and at-risk surgical population

SECONDARY OUTCOMES:
Conventional measure of metabolic equivalents (METS) | 0-1 day
  If conventional measures of METS (subjective METS, Duke Activity Status Index) compare favorably to the SHAPE testing performance variables.
Perioperative Morbidity Survey | 0-30 days
  • If SHAPE™ performance variables predict a higher risk of postoperative morbidity after surgery using the Postoperative Operative Morbidity Survey (POMS), a short-term measure of postoperative morbidity after major elective surgery.
Major postoperative outcomes | 0-30 days
  • If SHAPE™ performance variables predict a higher risk of postoperative major morbidity as measured by traditional major 30-day complications (myocardial infarction, stroke, atrial fibrillation, surgical site infection, postoperative pulmonary complications)

CONTACTS AND LOCATIONS:
Overall Officials: Zyad J Carr, M.D., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Variable description, values and deidentified patient physiological data.

REFERENCES:
- [Background] Ohnishi H, Inaba H, Mochizuki H, Kosuzume H. Mechanism of action of AC-1370 on phagocyte functions. Antimicrob Agents Chemother. 1984 Jan;25(1):88-92. doi: 10.1128/AAC.25.1.88. PMID 6703687
- [Background] Bennett H, Parfitt G, Davison K, Eston R. Validity of Submaximal Step Tests to Estimate Maximal Oxygen Uptake in Healthy Adults. Sports Med. 2016 May;46(5):737-50. doi: 10.1007/s40279-015-0445-1. PMID 26670455
- [Background] Bernstein EJ, Mandl LA, Gordon JK, Spiera RF, Horn EM. Submaximal heart and pulmonary evaluation: a novel noninvasive test to identify pulmonary hypertension in patients with systemic sclerosis. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1713-8. doi: 10.1002/acr.22051. PMID 23740875
- [Background] Bohannon RW, Crouch RH. Two-Minute Step Test of Exercise Capacity: Systematic Review of Procedures, Performance, and Clinimetric Properties. J Geriatr Phys Ther. 2019 Apr/Jun;42(2):105-112. doi: 10.1519/JPT.0000000000000164. PMID 29210933
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Cole CR, Blackstone EH, Pashkow FJ, Snader CE, Lauer MS. Heart-rate recovery immediately after exercise as a predictor of mortality. N Engl J Med. 1999 Oct 28;341(18):1351-7. doi: 10.1056/NEJM199910283411804. PMID 10536127
- [Background] Devereaux PJ, Goldman L, Cook DJ, Gilbert K, Leslie K, Guyatt GH. Perioperative cardiac events in patients undergoing noncardiac surgery: a review of the magnitude of the problem, the pathophysiology of the events and methods to estimate and communicate risk. CMAJ. 2005 Sep 13;173(6):627-34. doi: 10.1503/cmaj.050011. PMID 16157727
- [Background] Ferguson M, Shulman M. Cardiopulmonary Exercise Testing and Other Tests of Functional Capacity. Curr Anesthesiol Rep. 2022;12(1):26-33. doi: 10.1007/s40140-021-00499-6. Epub 2021 Nov 20. PMID 34840532
- [Background] Gerson MC, Hurst JM, Hertzberg VS, Baughman R, Rouan GW, Ellis K. Prediction of cardiac and pulmonary complications related to elective abdominal and noncardiac thoracic surgery in geriatric patients. Am J Med. 1990 Feb;88(2):101-7. doi: 10.1016/0002-9343(90)90456-n. PMID 2301435
- [Background] Grocott MP, Browne JP, Van der Meulen J, Matejowsky C, Mutch M, Hamilton MA, Levett DZ, Emberton M, Haddad FS, Mythen MG. The Postoperative Morbidity Survey was validated and used to describe morbidity after major surgery. J Clin Epidemiol. 2007 Sep;60(9):919-28. doi: 10.1016/j.jclinepi.2006.12.003. Epub 2007 May 7. PMID 17689808
- [Background] Hansen D, Jacobs N, Thijs H, Dendale P, Claes N. Validation of a single-stage fixed-rate step test for the prediction of maximal oxygen uptake in healthy adults. Clin Physiol Funct Imaging. 2016 Sep;36(5):401-6. doi: 10.1111/cpf.12243. Epub 2015 Jun 5. PMID 26046474
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Kallianos A, Rapti A, Tsimpoukis S, Charpidou A, Dannos I, Kainis E, Syrigos K. Cardiopulmonary exercise testing (CPET) as preoperative test before lung resection. In Vivo. 2014 Nov-Dec;28(6):1013-20. PMID 25398794
- [Background] Khatri V, Neal JE, Burger CD, Lee AS. Prognostication in Pulmonary Arterial Hypertension with Submaximal Exercise Testing. Diseases. 2015 Feb 6;3(1):15-23. doi: 10.3390/diseases3010015. PMID 28943605
- [Derived] Carr ZJ, Charchaflieh J, Brenes-Bastos A, He H, Lin HM, Jankelovits A, Gu E, Zafar J, Ghali F, Tan WS, Heerdt P. Preoperative submaximal cardiopulmonary exercise testing and its association with early postoperative complications. BJA Open. 2025 Apr 24;14:100407. doi: 10.1016/j.bjao.2025.100407. eCollection 2025 Jun. PMID 40421445
- [Derived] Carr ZJ, Agarkov D, Li J, Charchaflieh J, Brenes-Bastos A, Freund J, Zafar J, Schonberger RB, Heerdt P. Implementation of Brief Submaximal Cardiopulmonary Testing in a High-Volume Presurgical Evaluation Clinic: Feasibility Cohort Study. JMIR Perioper Med. 2025 Feb 17;8:e65805. doi: 10.2196/65805. PMID 39773953